CLINICAL TRIAL: NCT01753791
Title: A Phase 1, Dose Expansion Of A Within-cohort, Randomized, Double-blind, Third-party Open, Placebo-controlled, Single-and Multiple-dose Escalation Study To Evaluate Safety, Tolerability, And Pharmacokinetics Of Pf-06473871 In Normal Healthy Adults
Brief Title: Study To Evaluate Safety, Tolerability, And Pharmacokinetics Of PF-06473871 In Normal Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: B5301002; 2012-003797-13 (EudraCT Number)
Record Dates: First submitted 2012-11-20; First posted 2012-12-20 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Drug: 80 mg PF-06473871
- Cohort 2 (Experimental)
  Interventions: Drug: 160 mg PF-06473871
- Cohort 3 (Experimental)
  Interventions: Drug: 320 mg PF-06473871
- Cohort 4 (Experimental)
  Interventions: Drug: 480 mg PF-06473871

INTERVENTIONS:
Drug: 80 mg PF-06473871 — 80 mg of PF-06473871 or placebo
  Arms: Cohort 1
Drug: 160 mg PF-06473871 — 160 mg of PF-06473871 or placebo
  Arms: Cohort 2
Drug: 320 mg PF-06473871 — 320 mg of PF-06473871 or placebo
  Arms: Cohort 3
Drug: 480 mg PF-06473871 — 480 mg of PF-06473871 or placebo
  Arms: Cohort 4

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of PF-06473871 in normal healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or females between the ages of 18 and 55 years inclusive

Exclusion Criteria:

* Currently pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events | 6 weeks
  will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of subjects
ECGs | 6 weeks
  will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of subjects
Blood pressure | 6 weeks
  will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of subjects
pulse rate | 6 weeks
  will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of subjects
Injection siter reaction | 6 weeks
  The number and percentage of subjects that experienced injection site reactions will be analyzed.
number of subjects with adverse events | 6 weeks
  will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of subjects
severity of adverse events | 6 weeks
  will be reviewed and summarized on an ongoing basis during the study to evaluate the safety of subjects

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 6 weeks
Area under the Concentration-Time Curve (AUC) | 6 weeks
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Maximum Observed Plasma Concentration (Cmax) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5301002&StudyName=Study%20To%20Evaluate%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetics%20Of%20PF-06473871%20In%20Normal%20healthy%20Adults%20